CLINICAL TRIAL: NCT05186792
Title: Are Mycoplasma Species Associated With Disease in the Genitourinary System of Male and Female Patients Attending Sexual Health Clinics or Are They Bacterial Commensals?
Brief Title: Mycoplasma Species and the Genitourinary System
Status: Completed | Type: Observational
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: CT 253889
Record Dates: First submitted 2019-12-16; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2019-12

CONDITIONS: Sexually Transmitted Diseases, Bacterial
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- myco well participants: Retrospective analysis of patient records. No new patients recruited.
  Interventions: Other: Test:mycoplasma

INTERVENTIONS:
Other: Test:mycoplasma — Retrospective analysis of records of recruits to a previous mycoplasma study.

SUMMARY:
The purpose of this study is to determine if the presence of Mycoplasma hominis bacteria is associated with Bacterial vaginosis (BV), non-gonococcal urethritis (NGU) or vaginitis in patients attending sexual health clinic. Patients were participants of the MYCO WELL D-ONE study. Ethics for this follow-on pathway-to-portfolio study (IRAS:253889) is now approved by NRES and HCRW.

The important primary aim of this study is to determine if Mycoplasma hominis (M.hominis) is associated with BV, NGU and vaginitis in the genitourinary system of patients or if they are bacterial commensals. This is important proof of concept work. The secondary aim for this research is to determine if there are clinical and social parameters that are associated with Mycoplasma infection.

Preliminary analysis of 100 patients yielded pilot data suggesting M.hominis is strongly associated with BV, NGU and vaginitis. We aim to consolidate these findings by expansion to 1000 patients from our completed MYCOWELL D-ONE study.

DETAILED DESCRIPTION:
The clinical study site is The Department of Sexual Health, Dewi Sant Hospital, Cwm Taf University Health Board. This study will retrospectively examine the clinical notes of consented participants (IRAS project ID:253889) in the MYCO WELL D-ONE study (IRAS project ID:230693).

Notes will be identified by the sexual health clinic number. The clinic proforma records the following parameters:

1. Gender the patient identifies with
2. Age of the patient when the MYCO WELL D-ONE study sample collected
3. Symptoms and signs that were recorded in the patient notes e.g. BV/NGU
4. Previous sexually transmitted infections diagnosed
5. Drug history
6. Treatments the patient received
7. Sexual history e.g. type of sexual activity On completion, he parameters associated with positive M.hominis result; bacteria load quantification/antimicrobial resistance) and statistical analysis will be examined as below. I Statistical analysis This will be performed on anonymised data. The primary outcome measure of this study is to determine if M.hominis is associated with BV, NGU and vaginitis in the genitourinary system of patients or if it is a bacterial commensal. The secondary outcome for this research is to determine if there are clinical and social parameters that are associated with M.hominis infection.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active participants aged 18 to 100 years
* Participants can give informed consent in writing.

Exclusion Criteria:

* Patients who have been sexually assault.
* Participants who cannot give informed consent in writing.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are sexually active and attending a walk-in sexual health clinic in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
M. hominis and disease | 6 months
  Number of symptomatic participants with Mycoplasma infections

SECONDARY OUTCOMES:
M.hominis and drug use | 6 months
  Number of patients with Mycoplasma infection and drug use
M.hominis and number of sexual contacts | 6 months
  Number of patients with Mycoplasma infection who have more than 2 sexual partners in 3 months
M.hominis and miscarriage | 6 months
  Number of patients with Mycoplasma infection who have a history of miscarriage
M.hominis and abortion | 6 months
  Number of patients with Mycoplasma infection who have a history of abortion in the last 5 years
M.hominis and anal sex | 6 months
  Number of patients with Mycoplasma infection who perform anal sex
M.hominis and unprotected sex | 6 months
  Number of patients with Mycoplasma infection who have sex without condom use
M.hominis and contraception | 6 months
  Number of patients with Mycoplasma infection while taking hormonal contraception
M.hominis and men who have sex with men | 6 months
  Number of patients with Mycoplasma infection and are men that have sex with men
M.hominis and commercial sex workers | 6 months
  Number of patients with Mycoplasma infection who have sex with commercial sex workers
M.hominis and chemsex | 6 months
  Number of patients with Mycoplasma infection who have chemsex

CONTACTS AND LOCATIONS:
Locations (1):
- Cwm Taf Morgannwg University Health board, Pontypridd, United Kingdom

IPD SHARING:
Plan to Share IPD: No